CLINICAL TRIAL: NCT04257747
Title: Qualitative and Quantitative Evaluation of Vascular Flows of Radial, Ulnar and Interdigital Arterial Trees Under Normal and Pathological Conditions by 3 Tesla MRI
Acronym: FLOWHAND
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Collaborators: Hôpital Edouard Herriot (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: PI2019_843_0077
Record Dates: First submitted 2020-02-04; First posted 2020-02-06 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Magnetic Resonance Imaging; Vascular Complications; Transplantation; Radial Artery
Keywords: vascularized composite allotransplantation; hand allotransplantation; radial forearm flap; magnetic resonance imaging; flow MRI; radial artery; ulnar artery

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Healthy volunteers (Sham Comparator)
  Interventions: Other: MRI acquisitions; Other: Doppler ultrasound procedure
- patients requiring radial forearm flap reconstruction (Active Comparator)
  Interventions: Other: MRI acquisitions; Other: Doppler ultrasound procedure
- patients having received hand allotransplantation (Experimental)
  Interventions: Other: MRI acquisitions; Other: Doppler ultrasound procedure

INTERVENTIONS:
Other: MRI acquisitions — MRI acquisitions will be performed on the ACHIEVA 3T TX DStream Philips® Research MRI of the GIE Faire Faces.
Other: Doppler ultrasound procedure — The Doppler ultrasound procedure will be conducted in the traditional way in the Vascular Medicine Department of the Amiens-Picardie University Hospital

SUMMARY:
Allotransplants of vascularized composite tissues are subject to chronic vascular rejection, which can lead to graft loss. Currently, no imaging technique allows a reproducible quantitative exploration of the arterial trees of the hand, and therefore a satisfactory monitoring of transplants. Since 2014, flow MRI has been applied to the analysis of small-calibre arteries by the Image Processing Team at the Amiens-Picardie University Hospital. Between 2015 and 2017, several acquisitions were made in 3 patients who received facial allotransplantation, and the team recently developed a flow MRI protocol dedicated to the study of arterial trees in the hand.

The main objective is to measure vascular flows of radial, ulnar and interdigital arterial trees in normal (healthy volunteers) and pathological situations (patients with radial forearm flap reconstruction and patients with hand allotransplantation) using the specifically developed flow MRI protocol.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥ 18 years old)
* patients who has received appropriate information and provided informed consent
* patients benefiting from social security insurance
* patients with no contraindications to magnetic resonance imaging
* healthy volunteer or patient requiring radial forearm flap reconstruction or having received hand allotransplantation.

Exclusion Criteria:

* Person with a contraindication to MRI
* pregnant or breastfeeding woman
* minors (< 18 years)
* person under guardianship or deprived of liberty by a judicial or administrative decision
* person with upper limb arteriopathy with the exception of the hand transplant patients group.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Variation of radial vascular flows between healthy volunteers and patients with forearm flap reconstruction | day 0
  Radial vascular flows between healthy volunteers and patients with forearm flap reconstruction will be determined by using the specifically developed flow MRI protocol
Variation of ulnar artery vascular flows between healthy volunteers and patients with forearm flap reconstruction | day 0
  Ulnar artery vascular flows between healthy volunteers and patients with forearm flap reconstruction will be determined by using the specifically developed flow MRI protocol
Variation of interdigital arterial tree vascular flows between healthy volunteers and patients with forearm flap reconstruction | day 0
  Interdigital arterial tree vascular flows between healthy volunteers and patients with forearm flap reconstruction will be determined by using the specifically developed flow MRI protocol
Variation of radial vascular flows between healthy volunteers and patients with hand allotransplantation | day 0
  Radial vascular flows between healthy volunteers and patients with hand allotransplantation will be determined by using the specifically developed flow MRI protocol
Variation of ulnar artery vascular flows between healthy volunteers and patients with hand allotransplantation | day 0
  Ulnar artery vascular flows between healthy volunteers and patients with hand allotransplantation will be determined by using the specifically developed flow MRI protocol
Variation of interdigital arterial tree vascular flows between healthy volunteers and patients with hand allotransplantation | day 0
  Interdigital arterial tree vascular flows between healthy volunteers and patients with hand allotransplantation will be determined by using the specifically developed flow MRI protocol

CONTACTS AND LOCATIONS:
Overall Officials: Stéphanie Dakpe, MD, Principal Investigator — CHU Amiens; Jérémie Bettoni, MD, Principal Investigator — CHU Amiens; Olivier Baledent, MD, Principal Investigator — CHU Amiens; Marie-Antoinette Sevestre-Pietri, Pr, Principal Investigator — CHU Amiens; Emmanuel Morelon, Pr, Principal Investigator — Hopital Edouard Herriot; Palmira Petruzzo, MD, Principal Investigator — Hopital Edouard Herriot
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No